CLINICAL TRIAL: NCT00582686
Title: Prospective Comparison of Open Reduction Internal Fixation of Calcaneus Fractures With and Without Tricortical Iliac Crest Bone Grafting
Brief Title: Open Reduction Internal Fixation of Calcaneus Fractures With and Without Bone Graft
Acronym: CALCANEUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F990923008
Record Dates: First submitted 2007-12-20; First posted 2007-12-28 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Calcaneus Fractures
Keywords: Calcaneus Fractures; Iliac Crest Bone Grafting; Open Reduction & Internal Fixation
MeSH Terms: interventions — Bone Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ORIF with Bone Grafting (Active Comparator): This study will be designed as a randomized, prospective, blinded evaluation of patients who have sustained an intra-articular calcaneous fracture that would require open reduction with internal fixation as the preferred method of treatment. Group A will be made up of patients that undergo ORIF and Tricortical iliac crest bone grafting.
  Interventions: Procedure: ORIF of Calcaneus with bone grafting
- ORIF without Bone Grafting (Active Comparator): This study will be designed as a randomized, prospective, blinded evaluation of patients who have sustained an intra-articular calcaneous fracture that would require open reduction with internal fixation as the preferred method of treatment. Group B will consist of patients that undergo open reduction with internal fixation without bone grafting
  Interventions: Procedure: ORIF of Calcaneus without bone grafting

INTERVENTIONS:
Procedure: ORIF of Calcaneus with bone grafting — The calcaneus fracture will be surgically repaired with open reduction and internal fixation (ORIF) and Tricortical Iliac Crest bone grafting
  Arms: ORIF with Bone Grafting
Procedure: ORIF of Calcaneus without bone grafting — The calcaneus fracture will be surgically repaired with open reduction and internal fixation (ORIF) (no bone grafting)
  Arms: ORIF without Bone Grafting

SUMMARY:
The purpose of this study is to compare patient functional outcomes for surgical fixation of calcaneus fractures with and without tricortical iliac crest bone grafting

DETAILED DESCRIPTION:
This study was designed as a randomized, prospective evaluation of patients who have sustained an intra-articular calcaneus fracture that requires open reduction with internal fixation as the preferred method of treatment. Patients who desire to participate in this study will be randomized into one of two groups. Group A will be made up of patients that undergo open reduction with internal fixation and Tricortical iliac crest bone grafting. Group B will consist of patients that undergo open reduction with internal fixation without bone grafting. All other surgical techniques and management of the fracture and patient will remain unchanged.

ELIGIBILITY:
Inclusion Criteria:

* intra-articular calcaneus fractures requiring open reduction and internal fixation
* Adult patient (19 years or older)
* Mental capacity to comply with post-operative regimen, evaluation and data collection

Exclusion Criteria:

* non-operative fractures for primary or secondary reasons
* prior surgery to the hindfoot of the involved lower extremity
* inability to comply with post-operative regimen, evaluation and data collection
* inability or unwillingness to give informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2000-05; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Union and healing of Calcaneus Fracture | 3 month to 12 month healing period

CONTACTS AND LOCATIONS:
Overall Officials: Rena L Stewart, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham, Orthopaedic Trauma, Birmingham, Alabama, United States